CLINICAL TRIAL: NCT03753178
Title: Role of Sensory Potentials and High-resolution Ultrasonography in Confirmation of Common Peroneal Mononeuropathy at the Fibular Neck
Brief Title: Sensory Potentials and Ultrasonography in Common Peroneal Mononeuropathy
Status: Completed | Type: Observational
Sponsor: rania sanad (Other Government)
Responsible Party: Sponsor-Investigator, rania sanad, Principal Investigator, Zagazig University
Organization: Zagazig University (Other Government)
Other Study IDs: ZU-IRB#4729\ 24-6-2016
Record Dates: First submitted 2018-11-14; First posted 2018-11-26 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Common Peroneal Neuropathy
Keywords: ultrasonography; Common peroneal electrophysiological evaluations; Common peroneal neuropathy
MeSH Terms: conditions — Peroneal Neuropathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients: 70 participants presented with clinical and motor electrophysiological evidence of common peroneal neuropathy at the fibular neck
- controls: 70 controls

SUMMARY:
Common peroneal mononeuropathy at the fibular neck (CPN) is one of the most frequent mononeuropathies of the lower extremities.

The common peroneal nerve sub serves sensation to the dorsum of the foot and toes. In CPN motor fibers of the deep peroneal nerve are more frequently affected than those of the superficial peroneal nerve. Fascicles of the deep branch of the common peroneal nerve are more anteriorly located and more vulnerable to injury than those of the superficial peroneal branch. The clinical and electrodiagnostic findings in CPN resemble the anatomical structure of the common peroneal nerve, indeed fibers for the deep peroneal nerve and the superficial peroneal nerve are bounded in separate fascicles along the course of the nerve.

Superficial peroneal nerve sensory potential (SPSP) should be performed to localize the site of injury.

Electrodiagnostic testing is used widely to evaluate the function of the common peroneal nerve. SPSP have been examined in CPN with conflicting results. A loss in amplitude of this response implies some axonal loss affecting either the common peroneal nerve or its superficial branch. Prominent axonal loss is the hallmark of most CPN lesions and suggested that abnormalities in sensory nerves mirror those in motor nerves.

Moreover, assessment of the structure of the common peroneal nerve is likely to improve the diagnostic yield" by using high-resolution ultrasonography. Ultrasound imaging is painless, does not expose the patient to radiation, and has several advantages compared with magnetic resonance imaging in the laboratory setting, including reduced cost, accessibility, ability to image the entire length of the nerve in a single study, and the ability to image both statically and dynamically.

This study was conducted to evaluate the superficial peroneal sensory potential and high-resolution ultrasonography role in confirmation of common peroneal mononeuropathy at the fibular neck.

DETAILED DESCRIPTION:
The current study is a case control study that was done in the period from January 2015 to January 2016. The study included 70 participants presented with clinical and electrophysiological evidence of common peroneal neuropathy at the fibular neck (CPN) attending to Zagazig University Hospitals (Neurology, Rheumatology& Rehabilitation, and Orthopedic departments) and insurance hospitals of Sharkia governorate (47 male and 23 female). Their age (mean ± SD/years) was 40.4± 12.9, the duration between the onset of symptom and enrollment in the study ranged between 21 days to 6 months. Seventy (45 males and 25 females) apparently healthy volunteers were included as controls, and their age (mean ± SD/ years) was 41.3 ± 11.8. They were selected from the persons attending to blood bank for blood donation.

All participants included in the present study are subjected to:

1. Full history taking.
2. Thorough clinical and neurological examination.
3. Routine laboratories tests for exclusion of other systemic affection like diabetes mellitus, renal or hepatic failure.
4. Electrodiagnostic studies

   All tests were done in the same room, at the time of clinical diagnosis using a Nicolet Viking Quest cart electrodiagnostic system. Lower extremity temperature was maintained at or above 30º C at time of examination. The electrophysiological studies included the following:

   A-Motor nerve conduction studies:

   Motor conduction study of the common peroneal nerve (ankle-fibular neck -popliteal fossa), tibial motor nerve conduction study were performed with surface disc recording electrodes for the affected limb and the contralateral limb in all subjects. Evaluations of both upper limbs were added to exclude more wide lesions if suspected.

   Common peroneal CMAPs were recorded over extensor digitorum brevis and tibialis anterior.

   Investigators considered that the lesion is axonal via axonal loss estimation:

   Axonal loss of the motor branch of the common peroneal nerve was estimated by comparing the CMAP amplitude recorded from the extensor digitorum brevis on the affected and contralateral sides.

   An estimate of EDB axonal loss was obtained from the formula (U -A)/U ×100 U : (extensor digitorum brevis response amplitude from the unaffected side).

   A : (extensor digitorum brevis response amplitude from the affected side).

   Categorization based on the motor estimated axonal loss as follow:

   No loss: (<50%). Mild to moderate loss: (50-75%). Severe loss: (>75%).

   B- Sensory nerve conduction studies:

   Antidromic evaluation of the superficial peroneal nerve sensory potential (SPSP) at the ankle was studied with surface stimulating and recording electrodes on the affected limb and the contralateral limb in all subjects. The site of stimulation was just anterior to the edge of the shaft of the fibula and 14 cm proximal to the active ankle electrode. The active recording electrode was placed midway between the edge of the tibia and the tip of the lateral malleolus or 3 cm proximal to the bimalleolar line. The reference recording electrode was placed 3 cm distal to the active electrode.

   SPSP was considered affected when any one of the following is detected :
   * No constant wave forms could be detected.
   * SPSP amplitudes < 5 μv or < 50% of the contra lateral side.
   * Increased peak latency ≥ 4.4 ms (based on standard distance of 14 cm).

   C-Electromyographic study (EMG) was carried out using concentric needle in the following muscles: extensor digitorum brevis (EDB), tibialis anterior, peroneus longus, tibialis posterior, extensor halucis longus, short head of biceps femoris, vastus lateralis, medial head of gastrocnemius, iliacus, gluteus medius, tensor fascia lata and Paraspinal muscles. Concentric needle EMG was performed in all patients. Spontaneous and voluntary motor unit activity was assessed.
5. Radiological examination:

A) Ultrasonographic assessment of participants:

Ultrasonographic examination by radiologist was conducted with a General Electric Logiq 7 Pro machine (GE Healthcare, Chalfont St Giles, England), using a 5- to 12-MHz linear array transducer. The cross sectional area (CSA) of the common peroneal nerve was determined within the echogenic rim surrounding the nerve at the level of the fibular neck with the probe perpendicular to the main nerve course in the transverse and longitudinal plane. The sonographic measurements were done on the same day or within 1 week after the electrodiagnostic studies.

The radiologist was blinded to the participants' electrophysiological study data. However, the radiologist was aware of the clinical and electrophysiological suspicion for common peroneal neuropathy.

Authors of the present study considered that common peroneal nerve is affected by the sonographic measurements if the value of CSA of the common peroneal nerve at the fibular neck was >11 mm2 according to the study control group.

B) Plain radiographs were done to detect the underlying traumatic injuries, such as a proximal fibular head fracture or osseous tumors, or in assessing the severity of angular deformities about the knee. Lumbosacral plain X ray or MRI were done only if needed to rule lumbosacral affection.

ELIGIBILITY:
Inclusion Criteria:

* Participants were eligible for inclusion in the study if they had clinical and motor electrophysiological evidence suggesting common peroneal mononeuropathy at the fibular neck

Clinical evidence of common peroneal mononeuropathy at the fibular neck:

* Numbness of the antero lateral aspect of the lower limb from about midway between the knee and the ankle, most of the dorsal aspect of the foot and toes and the web space between the first and second toes.
* Weakness of the leg muscles innervated by the peroneal nerve. The strength of the tibialis anterior (TA), extensor hallucislongus (EHL), and peroneius longus muscles was tested using the Medical Research Council (MRC) rating scale.

Electrophysiological Motor localizing evidence of common peroneal mononeuropathy at the fibular neck:

Peroneal motor nerve conduction velocity decrement ≥10 m/s across the fibular neck segment; or focal conduction block, defined as compound motor action potential (CMAP) amplitude and area reduction ≥ 50% across the fibular neck segment.

Exclusion Criteria:

* Participants were excluded if any of the following was detected:

  * Historical or clinical signs suggesting coexisting neurological conditions (e.g. polyneuropathy and motor neuropathy).
  * Foot drop with symptoms, signs or radiological findings of L5 radiculopathy in association with CPN.
  * Symptoms or signs suggesting systemic clinical illness like diabetes mellitus, renal failure, and hepatic failure.
  * Previous surgery for peroneal nerve.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 70 (47 male and 23 female) patients presented with clinical and electrophysiological evidence of common peroneal neuropathy at the fibular neck attending to Zagazig University Hospitals and insurance hospitals of Sharkia governorate. Their age (mean ± SD/years) was 40.4± 12.9, the duration between the onset of symptom and enrollment in the study ranged between 21 days to 6 months. Seventy (45 males and 25 females) apparently healthy volunteers were included as controls, and their age (mean ± SD/ years) was 41.3 ± 11.8.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-01-31 (Actual); Study Completion 2016-01-31 (Actual)

PRIMARY OUTCOMES:
is measuring the common peroneal nerve electrophysiological studies | two week
  measuring the common peroneal nerve senseromotor electrophysiological studies
is measuring the common peroneal nerve Ultrasonographical studies | 1 week
  measuring the common peroneal nerve Ultrasonographical cross sectional area

IPD SHARING:
Plan to Share IPD: Yes
Study is to be shared with other researchers.
Supporting Information: Study Protocol, SAP
Time Frame: the data will become available ( for six months) after publishing it in the Egyptian Journal of Neurology, Psychiatry and Neurosurgery
URL: http://ejnpn.springeropen.com